CLINICAL TRIAL: NCT04096196
Title: Safe City: a Game-based Educational Approach to Promote Child Safety Knowledge and Behaviours
Brief Title: A Game-based Educational Approach to Promote Child Safety Knowledge and Behaviours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SC2019HK
Record Dates: First submitted 2019-09-13; First posted 2019-09-19 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2022-05

CONDITIONS: Injuries; Knowledge, Attitudes, Practice
MeSH Terms: conditions — Wounds and Injuries; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game intervention group (Experimental): Participants assigned to the intervention group will be given a manual containing instructions to play the Safe City game. A research assistant will provide a briefing session on the game in each participating school. A unique username and password set will be created for each user to log in the game. This login information will be provided to the student participants in a sealed envelope after the briefing session. The participants will be instructed to play the game as many times as desired within a 4-week time frame. The players ranked in the top 20 will receive a reward in the form of book coupon after the intervention ends.
  Interventions: Behavioral: Safe City game
- Health education ("control") group (Active Comparator): All students in the health education group will receive a comprehensive package on safety information. The information package includes both printed and electronic promotional materials regarding safety and a comprehensive list of relevant website and information sources. The information from these relevant websites and information sources are similar to those used in setting the safety case scenarios for the Safe City game. As a result, both intervention arms will have comparable accessibility to safety-related information and the major contrast between the two groups will be the method of presentation (game-based learning vs traditional health promotion approach, i.e. unidirectional information package).
  Interventions: Other: Health education

INTERVENTIONS:
Behavioral: Safe City game — The game intervention uses a game-based learning approach to teach players how to recognize and remove injury hazards from different homes and sports areas. It also highlights the need to pay attention to traffic and safety facilities to prevent injuries in a real-world environment. Players will create their own avatar to assume the duties of safety inspectors in the game. Point, level and reward systems will be included to increase player motivation to engage in the game.
  Arms: Game intervention group
Other: Health education — All students in the health education group will receive a comprehensive package on safety information. The information package includes both printed and electronic promotional materials regarding safety and a comprehensive list of relevant website and information sources. The information from these relevant websites and information sources are similar to those used in setting the safety case scenarios for the Safe City game. As a result, both intervention arms will have comparable accessibility to safety-related information and the major contrast between the two groups will be the method of presentation (game-based learning vs traditional health promotion approach, i.e. unidirectional information package).
  Arms: Health education ("control") group

SUMMARY:
The project will design and develop a game for teaching safety as a way to reduce childhood injury. To evaluate the effectiveness of the designed game, a randomized controlled trial (RCT) following the CONSORT RCT guidelines will be conducted. All students in Primary 4-6 (equivalent to US Grades 4-6) from the participating school will be invited to join the trial, which will be then randomized into the game or health education group. All students in the game group will be invited to play the designed game with instructions provided, while those in health education group will receive a comprehensive package on safety information. The intervention will last 4 weeks, with the safety knowledge and behaviours, and psychosocial difficulties of the participants being assessed before and 1 and 3 months after the intervention. The effectiveness of the intervention in achieving the proposed targets will be estimated using linear mixed models.

DETAILED DESCRIPTION:
To evaluate the effectiveness of the Safe City game, a randomized controlled trial (RCT) following the CONSORT RCT guidelines will be conducted.The evaluation will therefore be conducted in four school districts. An invitation will be sent to each selected school. After the school principal agrees to join the trial, informed written consents will be obtained from parents of the participating students by our research staff before randomization. The participant recruitment and randomization process will be independently carried out by different research assistants. Outcome assessors will be blinded to the allocation of participants in each group.

All consenting student participants, before intervention, will be asked to complete a questionnaire on basic socio-demographics. The intervention will last 4 weeks. Their safety knowledge and behaviours, HRQOL and psychosocial difficulties will be assessed before and 1 and 3 months after the intervention.

Game ("intervention") group The Safe City game intervention uses a game-based learning approach to teach players how to recognize and remove injury hazards from different homes and sports areas. It also highlights the need to pay attention to traffic and safety facilities to prevent injuries in a real-world environment. Players will create their own avatar to assume the duties of safety inspectors in the game. Point, level and reward systems will be included to increase player motivation to engage in the game.

Participants assigned to the intervention group will be given a manual containing instructions to play the Safe City game. A research assistant will provide a briefing session on the game in each participating school. A unique username and password set will be created for each user to log in the game. This login information will be provided to the student participants in a sealed envelope after the briefing session. The participants will be instructed to play the game as many times as desired within a 4-week timeframe. The players ranked in the top 20 will receive a reward in the form of book coupon after the intervention ends.

Health education ("control") group All students in the health education group will receive a comprehensive package on safety information. The information package includes both printed and electronic promotional materials regarding safety and a comprehensive list of relevant website and information sources. The information from these relevant websites and information sources are similar to those used in setting the safety case scenarios for the Safe City game. As a result, both intervention arms will have comparable accessibility to safety-related information and the major contrast between the two groups will be the method of presentation (game-based learning vs traditional health promotion approach, i.e. unidirectional information package).

ELIGIBILITY:
Inclusion Criteria:

Hong Kong Chinese children studying in Primary 4 to 6 Enrolling in non-special, local (non-international) primary schools in the 4 selected districts (Kwai Tsing, North, Sham Shui Po, and Tai Po)

Exclusion Criteria:

Non-Chinese speaking subjects. Non-consenting subjects.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 340 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Changes from baseline safety knowledge at 1 month | At baseline and 1 and 3 months after the intervention
  Child safety knowledge will be measured by different items adopted from the existing literature and questionnaires under the three contexts: home safety, road safety, and sports-related safety. Child participants will be asked to indicate their level of involvement in the said behaviour on a 5-point Likert scale ranging from "Never" to "Very Often", or their agreement on the given statement based upon their own safety knowledge on a 4-point Likert scale ranging from "Strongly disagree" to "Strongly agree".
Changes from baseline safety knowledge at 3 months | At baseline and 1 and 3 months after the intervention
  Child safety knowledge will be measured by different items adopted from the existing literature and questionnaires under the three contexts: home safety, road safety, and sports-related safety. Child participants will be asked to indicate their level of involvement in the said behaviour on a 5-point Likert scale ranging from "Never" to "Very Often", or their agreement on the given statement based upon their own safety knowledge on a 4-point Likert scale ranging from "Strongly disagree" to "Strongly agree".
Changes from baseline safety behaviours at 1 month | At baseline and 1 and 3 months after the intervention
  Child safety behaviours will be measured by different items adopted from the existing literature and questionnaires under the three contexts: home safety, road safety, and sports-related safety. Child participants will be asked to indicate their level of involvement in the said behaviour on a 5-point Likert scale ranging from "Never" to "Very Often", or their agreement on the given statement based upon their own safety knowledge on a 4-point Likert scale ranging from "Strongly disagree" to "Strongly agree".
Changes from baseline safety behaviours at 3 months | At baseline and 1 and 3 months after the intervention
  Child safety behaviours will be measured by different items adopted from the existing literature and questionnaires under the three contexts: home safety, road safety, and sports-related safety. Child participants will be asked to indicate their level of involvement in the said behaviour on a 5-point Likert scale ranging from "Never" to "Very Often", or their agreement on the given statement based upon their own safety knowledge on a 4-point Likert scale ranging from "Strongly disagree" to "Strongly agree".

SECONDARY OUTCOMES:
Changes from baseline child generic quality of life at 1 month | At baseline and 1 and 3 months after the intervention
  Child generic quality of life will be measured by the Chinese version of the PedsQL Generic Core Scales (Child-Self Report version) which has four subscales with a total of 23 items measuring the physical, emotional, social, and school functioning of the children. Each item is rated on a 5-point scale from 0=never to 4=almost always. A higher score indicates better functioning.
Changes from baseline child generic quality of life at 3 months | At baseline and 1 and 3 months after the intervention
  Child generic quality of life will be measured by the Chinese version of the PedsQL Generic Core Scales (Child-Self Report version) which has four subscales with a total of 23 items measuring the physical, emotional, social, and school functioning of the children. Each item is rated on a 5-point scale from 0=never to 4=almost always. A higher score indicates better functioning.
Changes from baseline children behaviours at 1 month | At baseline and 1 and 3 months after the intervention
  Strength and Difficulties Questionnaire (SDQ) will be used to measure children's behaviour. The SDQ has five subscales, including emotional symptoms, conduct problems, peer relationship problems, hyperactivity/inattention, and prosocial behaviour. Each subscale has a score, and the first four subscales generate a total score of difficulties (20 items)
Changes from baseline children behaviours at 3 months | At baseline and 1 and 3 months after the intervention
  Strength and Difficulties Questionnaire (SDQ) will be used to measure children's behaviour. The SDQ has five subscales, including emotional symptoms, conduct problems, peer relationship problems, hyperactivity/inattention, and prosocial behaviour. Each subscale has a score, and the first four subscales generate a total score of difficulties (20 items)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Ip, MBBS, MPH, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong RS, Tung KTS, Ho FKW, Wong WHS, Chow CB, Chan KL, Fu KW, Ip P. Effect of a Mobile Game-Based Intervention to Enhance Child Safety: Randomized Controlled Trial. J Med Internet Res. 2024 Feb 14;26:e51908. doi: 10.2196/51908. PMID 38354042
- [Derived] Wong RS, Tung KT, Wong HT, Ho FK, Wong HS, Fu KW, Pong TC, Chan KL, Chow CB, Ip P. A Mobile Game (Safe City) Designed to Promote Children's Safety Knowledge and Behaviors: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Jun 12;9(6):e17756. doi: 10.2196/17756. PMID 32530436